CLINICAL TRIAL: NCT04949113
Title: Multicenter Phase 3 Trial Comparing Neoadjuvant Ipilimumab Plus Nivolumab Versus Standard Adjuvant Nivolumab in Macroscopic Stage III Melanoma - NADINA
Brief Title: Neoadjuvant Ipilimumab Plus Nivolumab Versus Standard Adjuvant Nivolumab in Macroscopic Stage III Melanoma
Acronym: NADINA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M21NDN; CA209-6FR (Other: BMS)
Record Dates: First submitted 2021-06-16; First posted 2021-07-02 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Malignant Melanoma Stage III
Keywords: Checkpoint inhibition; Checkpoint inhibitor; Immunotherapy; PD-1 inhibitor; CTLA-4 inhibitor; Ipilimumab; Nivolumab; Neoadjuvant; Adjuvant; Resectable melanoma; NADINA; M21NDN; Checkpoint blockade
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Open-label two-arm randomized phase 3 trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- A: Neoadjuvant (Experimental): 2 cycles of neoadjuvant ipilimumab (80mg) + nivolumab (240mg) every 3 weeks followed by a total lymph node dissection (TLND) and if applicable, resection of in-transit metastases.
  Patients with a pathologic partial or non-response in arm A will also receive adjuvant nivolumab 480 mg every 4 weeks 11 cycles. In case of BRAF V600E/K mutation-positivity, patients will be treated with adjuvant dabrafenib plus trametinib for 46 weeks instead.
  Interventions: Drug: Neoadjuvant ipilimumab + nivolumab
- B: Adjuvant (Active Comparator): Standard upfront total lymph node dissection (TLND) and if applicable, resection of in-transit metastases followed by 12 cycles adjuvant nivolumab 480 mg every 4 weeks
  Interventions: Drug: Adjuvant nivolumab

INTERVENTIONS:
Drug: Neoadjuvant ipilimumab + nivolumab — 2 cycles ipilimumab (80mg) + nivolumab (240mg) every 3 weeks followed by total lymph node dissection
  Other Names: Yervoy + Opdivo
  Arms: A: Neoadjuvant
Drug: Adjuvant nivolumab — Upfront total lymph node dissection followed by 12 cycles of nivolumab (480mg) every 4 weeks.
  Other Names: Opdivo
  Arms: B: Adjuvant

SUMMARY:
This is an international (Australia, Europe, and USA) open-label two-arm randomized phase 3 trial including 420 stage III (≤3 resectable in-transit metastases allowed) cutaneous or unknown primary melanoma patients. Patients will be randomized 1:1 to receive either 2 cycles of neoadjuvant ipilimumab 80 mg + nivolumab 240 mg every 3 weeks followed by a total lymph node dissection (TLND) and, if applicable, resection of in-transit metastases (arm A) versus standard upfront TLND +/- resection of in-transit metastases followed by 12 cycles adjuvant nivolumab 480 mg every 4 weeks (arm B). Patients with a pathologic partial or non-response in arm A will also receive adjuvant nivolumab 480 mg every 4 weeks for 46 weeks (11 cycles). In case of BRAF V600E/K mutation-positivity, patients from arm A with a pathologic partial or non-response (>10% viable tumor) will be treated with adjuvant dabrafenib plus trametinib for 46 weeks. Patients will be treated in the study in both arms until melanoma progression to irresectable stage III or stage IV disease, disease recurrence, unacceptable toxicity, subject withdrawal of consent or until end of study treatment.

An interim analysis will be performed after 60 events have occurred. The data safety monitory board (DSMB) will be ad hoc consulted when unexpected toxicities are reported. Patients will be followed by 12 weekly CT scans until end of year 3 and then until year 5 according to the institute's standards.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, at least 16 years of age;
* World Health Organization (WHO) Performance Status 0 or 1;
* Cytologically or histologically confirmed resectable stage III melanoma of cutaneous or unknown primary origin with one or more macroscopic lymph node metastases (clinical detectable), that can be biopsied and a maximum of 3 additional resectable in-transit metastases. A concurrent resectable primary melanoma is allowed. Clinical detectable lymph nodes are defined as either a palpable node, confirmed as melanoma by pathology, or a non-palpable but enlarged lymph node according to RECISTv1.1 (at least 15 mm in short axis), confirmed as melanoma by pathology, or a PET scan positive lymph node of any size confirmed as melanoma by pathology;
* No other malignancies, except adequately treated and with a cancer-related life-expectancy of more than 5 years;
* No prior immunotherapy targeting CTLA-4, PD-1 or PD-L1;
* No prior targeted therapy targeting BRAF and/or MEK;
* No immunosuppressive medications within 6 months prior study inclusion (steroids equivalent to prednisolone ≤10 mg are allowed);
* Screening laboratory values must meet the following criteria: WBC ≥2.0x109/L, neutrophils ≥1.5x109/L, platelets ≥100x109/L, hemoglobin ≥5.5 mmol/L, creatinine ≤1.5xupper limit of normal (ULN), AST ≤1.5x ULN, ALT ≤1.5x ULN, bilirubin ≤1.5x ULN (except for subjects with Gilbert syndrome who must have a total bilirubin <3.0 mg/dL);
* LDH level <1.5x ULN;
* Women of childbearing potential (WOCP) must use appropriate method(s) of contraception, i.e. methods with a failure rate of <1% per year when used consistently and correctly, to avoid pregnancy for 23 weeks post last ipilimumab + nivolumab infusion;
* Males who are sexually active with WOCP must use appropriate method(s) of contraception, i.e. methods with a failure rate of <1% per year when used consistently and correctly, to avoid pregnancy for 31 weeks post last ipilimumab + nivolumab infusion;
* Patient willing and able to understand the protocol requirements and comply with the treatment schedule, scheduled visits, electronic patient outcome reporting, tumor biopsies and extra blood withdrawal during screening and in case of recurrence, and other requirements of the study;
* Patient has signed the Informed Consent document.

Exclusion Criteria:

* Distantly metastasized melanoma;
* Uveal/ocular or mucosal melanoma;
* In-transit metastases only (without cytological or histological proven lymph node involvement)
* Subjects with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications. Subjects with resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, are permitted to enroll;
* Prior radiotherapy;
* Subjects will be excluded if they test positive for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus ribonucleic acid (HCV antibody), indicating acute or chronic infection. Subjects treated and being at least one year free from HCV are allowed to participate;
* Subjects will be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS);
* Subjects with history of allergy to study drug components or history of severe hypersensitivity reaction to monoclonal antibodies.
* Subjects with underlying medical conditions or active infection that, in the investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events;
* Women who are pregnant or breastfeeding;
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids >10 mg prednisolone daily equivalent;
* Use of other investigational drugs before study drug administration 30 days or 5 half-times before study inclusion;
* Psychological, familial, sociological, or geographical conditions that potentially hamper compliance with the study protocol and follow-up schedule; those conditions should be discussed with the subject before registration in the trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2028-12-19 (Estimated)

PRIMARY OUTCOMES:
Comparison of event-free survival (EFS) in the neoadjuvant and adjuvant group. | Analysis will be performed after 132 events, though not later than after 2 years follow-up of all patients.
  EFS is defined as time from randomization to melanoma progression (irresectable stage III or stage IV disease), melanoma recurrence, treatment-related death, or melanoma-related death, whichever occurs first. Occurrence of a new primary melanoma during treatment/follow-up is also regarded as an event. Presurgical resectable progression to stage III disease in arm A is not defined as an event, even as death to another reason than melanoma or the study treatment.

SECONDARY OUTCOMES:
Recurrence free survival (RFS) | Up to 5 years after randomization
  RFS is defined as time between date of surgery and date of melanoma recurrence, treatment-related death or melanoma-related death, whichever occurs first.
Distant metastases-free survival (DMFS) | Up to 5 years after randomization
  DMFS is defined as time between date of randomization and date of first distant metastasis, treatment-related death or melanoma-related death, whichever occurs first.
Overall survival (OS) | Up to 5 years after randomization
  OS is defined as time between date of randomization and date of death.
Pathologic response rate in the neoadjuvant arm and evaluation of association between pathologic response rate and RFS, DMFS and OS. | Up to 5 years after randomization
  The pathologic response rate will be categorized into pathologic complete response (pCR), near-pCR, major pathologic response (MPR), pathologic partial response (pPR), pathologic no response (pNR), according to International Neoadjuvant Melanoma Consortium (INMC) criteria.
Rate of immune-related adverse events | Up to 5 years after randomization
  Frequency of all grade and grade 3-5 treatment-related adverse events according to CTCAE 5.0.
Duration of immune-related adverse events | Up to 5 years after randomization
  Duration of all grade and grade 3-5 treatment-related adverse events according to CTCAE 5.0.
Description of type of immune-related adverse events | Up to 5 years after randomization
  Type of all grade and grade 3-5 treatment-related adverse events according to CTCAE 5.0.
Description of surgical morbidity | Up to 5 years after randomization
  Surgical complication rates according to Clavien-Dindo surgical classification.
Evaluation of health-related quality of life (HRQoL) in both treatment arms | Up to 5 years after randomization
  Quality of life as measured by EORTC Quality of Life Questionnaire-core 30 (QLQ C30). The QLQ-C30 is scored on 4 point Likert-scales: "Not at all", "A little", "Quite a bit", and "Very much." and is composed of both multi-item scales and single-item measures. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Evaluation of health-related quality of life (HRQoL) in both treatment arms | Up to 5 years after randomization
  Quality of life as measured by the Melanoma Subscale and Melanoma Surgery Subscale of Functional Assessment of Cancer Therapy - Melanoma (FACT-M). The FACT-M is scored on a 5 point Likert-scale: "Not at all", "A little bit", "Somewhat", "Quite a bit", and "Very much.". A Higher score represents higher Health Related Quality of Life (HRQoL).
Evaluation of health-related quality of life (HRQoL) in both treatment arms | Up to 5 years after randomization
  Quality of life as measured by the Cancer Worry Scale. The Cancer Worry Scale is scored on a 4 point Likert-scale: "Almost never", "Sometimes", "Often", and "Almost always". Higher scores indicate more worrying about cancer.
Evaluation of health-related quality of life (HRQoL) in both treatment arms | Up to 5 years after randomization
  Quality of life as measured by the Hospital Anxiety and Depression Scale (HADS) questionnaire. The HADS is a questionnaire that is scored on several 4 point Likert-scales. Higher score on the HADS questionnaire indicates more hospital-related anxiety and depression.
Evaluation of health-related quality of life (HRQoL) in both treatment arms | Up to 5 years after randomization
  Quality of life as measured by the 5-level EuroQOL-5D questionnaire (EQ-5D-5L).
Evaluation of health-related quality of life (HRQoL) in both treatment arms | Up to 5 years after randomization
  Quality of life as measured by an immunotherapy-specific questionnaire.
Evaluation of health-related quality of life (HRQoL) in both treatment arms | Up to 5 years after randomization
  Quality of life as measured by an assessment of work performance.
Evaluation of health-related quality of life (HRQoL) in both treatment arms | Up to 5 years after randomization
  Quality of life as measured by a questionnaire on sexual health.
Evaluation of health-related quality of life (HRQoL) in both treatment arms | Up to 5 years after randomization
  Quality of life as measured by the Amsterdam Cognition Scale.
Health technology assessments, consisting of a cost-effectiveness analysis comparing the neoadjuvant arm with the standard adjuvant arm | Up to 5 years after randomization
  Cost-effectiveness measured by an incremental cost-effectiveness ratio (ICER) (e.g., incremental cost per quality-adjusted life-year (QALY) gained).

CONTACTS AND LOCATIONS:
Overall Officials: Christian Blank, Prof, Study Chair — Medical oncologist/researcher; Georgina Long, Prof, Study Chair — Medical oncologist/researcher
Locations (24):
- United States (2):
  - The Angeles Clinic, Los Angeles, California
  - MD Anderson Cancer Center, Houston, Texas
- Australia (8):
  - Melanoma Institute Australia (MIA), Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane
  - Lake Macquarie Private Hospital, Gateshead
  - Alfred Health, Melbourne
  - Peter MacCallum Cancer Center, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Tasman Oncology, Southport
  - Westmead Hospital, Sydney
- Netherlands (14):
  - Netherlands Cancer Institute, Amsterdam, North Holland
  - Amsterdam University Medical Center - location VUmc, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Maxima Medisch Centrum, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Zuyderland Medisch Centrum, Heerlen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht
  - Isala Hospital, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blank CU, Lucas MW, Scolyer RA, van de Wiel BA, Menzies AM, Lopez-Yurda M, Hoeijmakers LL, Saw RPM, Lijnsvelt JM, Maher NG, Pulleman SM, Gonzalez M, Torres Acosta A, van Houdt WJ, Lo SN, Kuijpers AMJ, Spillane A, Klop WMC, Pennington TE, Zuur CL, Shannon KF, Seinstra BA, Rawson RV, Haanen JBAG, Ch'ng S, Naipal KAT, Stretch J, van Thienen JV, Rtshiladze MA, Wilgenhof S, Kapoor R, Meerveld-Eggink A, Grijpink-Ongering LG, van Akkooi ACJ, Reijers ILM, Gyorki DE, Grunhagen DJ, Speetjens FM, Vliek SB, Placzke J, Spain L, Stassen RC, Amini-Adle M, Lebbe C, Faries MB, Robert C, Ascierto PA, van Rijn R, van den Berkmortel FWPJ, Piersma D, van der Westhuizen A, Vreugdenhil G, Aarts MJB, Stevense-den Boer MAM, Atkinson V, Khattak M, Andrews MC, van den Eertwegh AJM, Boers-Sonderen MJ, Hospers GAP, Carlino MS, de Groot JB, Kapiteijn E, Suijkerbuijk KPM, Rutkowski P, Sandhu S, van der Veldt AAM, Long GV. Neoadjuvant Nivolumab and Ipilimumab in Resectable Stage III Melanoma. N Engl J Med. 2024 Nov 7;391(18):1696-1708. doi: 10.1056/NEJMoa2402604. Epub 2024 Jun 2. PMID 38828984
- [Derived] Long GV, Menzies AM, Scolyer RA. Neoadjuvant Checkpoint Immunotherapy and Melanoma: The Time Is Now. J Clin Oncol. 2023 Jun 10;41(17):3236-3248. doi: 10.1200/JCO.22.02575. Epub 2023 Apr 27. PMID 37104746